CLINICAL TRIAL: NCT03478410
Title: Role of Exosomes Derived From Epicardial Fat in Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Eilon Ram, Resident in cardiac surgery, Principal Investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHEBA-18-4516-ER-CTIL
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
Keywords: Epicardial fat
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Comparative study between patients with and without atrial fibrillation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atrial fibrillation (Other): An epicardial fat biopsy will be taken from patients with chronic atrial fibrillation or paroxysmal atrial fibrillation who undergo any cardiac surgery
  Interventions: Procedure: Epicardial fat biopsy
- Control (Other): An epicardial fat biopsy will be taken from patients without any history of atrial fibrillation who undergo any cardiac surgery
  Interventions: Procedure: Epicardial fat biopsy

INTERVENTIONS:
Procedure: Epicardial fat biopsy — A 1 cm (~0.5 g) of epicardial pat biopsy from the area of the pulmonary artery

SUMMARY:
Exosome plays an important role in the pathophysiology of the cardiovascular system. Since the field of cardiovascular exosome is still in its infancy, there are no available data regarding to its role in cardiac arrhythmias. The current study investigates the role of epicardial fat derived exosomes in patients who suffer from atrial fibrillation.

DETAILED DESCRIPTION:
Myocardial cells communication is mediated via direct cell to cell contact, cell to matrix interaction, long-range signals, electrical signals, and via extracellular chemical molecules (such as proteins, nucleotides, lipids and short peptides). Cell to cell communication can be achieved through direct contact (i.e. Gap junction, cell surface protein/protein interaction) or via secreted signaling molecules (i.e. hormones, neurotransmitters, cytokines). In the last few decades, a third intercellular communication mechanism has gained intense attention - extracellular vesicles that include: (1) apoptotic vesicles (1000-4000 nm), (2) microvesicles (100 nm - 1000 nm), and the smallest extracellular vesicles (3) exosomes (40-100 nm).

The exosomes are produced through the endosomal pathway and are able to carry cargo and transfer them to recipient cells, thus contributing to cell-to-cell communication. The exosomes cargo includes protein content, rRNA, tRNA, short DNA sequences, messenger RNA (mRNA) and microRNA (miRNA). The last two can change the gene expression within the target cells and by that affect myocardial cells.

Nowadays, it is known that in the cardiovascular system, exosome plays important roles in the pathophysiology of myocardial infarction (MI) and as an indicator for the damage and repair mechanisms post-acute MI (i.e. miR-126), in myocardial remodeling, and cardiac regeneration.

Since the field of cardiovascular exosome is still in its infancy, there are no available data regarding to its role in cardiac arrhythmias. Therefore, there is place to investigate the role of exosomes in patients who suffer from atrial fibrillation.

Some of the important issues to explore are: (1) Do the epicardial fat in patients with atrial fibrillation release quantitatively and qualitatively different exosomes than in patients without atrial fibrillation? (2) Can epicardial fat exosomes be a clinical biomarker for arrhythmias? (3) Can these exosomes be a target for the treatment and prevention of arrhythmias?

The current study will include patients who undergo any cardiac surgery and will give informed consent. An epicardial fat biopsy will be taken and cultured in a medium that contain M-199 medium, dexamethasone, gentamicin, and insulin for 9 days. The exosomes will be collected from the medium and analyzed.

The participants will be divided into two groups: (1) participants with atrial fibrillation, (2) participants who did not develop ever atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing an elective cardiac surgery

Exclusion Criteria:

* Undergoing a non-elective surgery
* Suffering from severe renal impairment prior to surgery (creatinine clearance <30 mL/min)
* Experienced hepatic dysfunction other than mild

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-01-21 (Actual); Primary Completion 2022-01-21 (Estimated); Study Completion 2022-01-21 (Estimated)

PRIMARY OUTCOMES:
Exosomes quantity excreted from the epicardial fat (nm) | 9 days
  The differences in the quantity of exosomes derived epicardial fat in patients with and without atrial fibrillation.
  The exosome isolation will be done by using ultra centrifuge for cells and cells debris removal.
  Then the exosomes will examined by the Malvern NanoSight device both for particle size and concentration measurement.

SECONDARY OUTCOMES:
Inflammatory cytokines secretion from epicardial fat | 9 days
  The differences in the Inflammatory cytokines secreted from epicardial fat in patients with and without atrial fibrillation.
  The investigators will detect the levels of cytokines and acute phase proteins such as IL1, IL2, IL6, IL8, IL10, IL12, CRP, VEGF, TNF-a, and TGF by Human Cytokine Array Kit.

CONTACTS AND LOCATIONS:
Overall Officials: Eilon Ram, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Results: The exosomes content in patients with and without atrial fibrillation